CLINICAL TRIAL: NCT06051981
Title: The Effect of Fluoride Varnish, Casein Phosphopeptide-Amorphous Calcium Phosphate, and Resin Infiltration in the Treatment of White Spot Lesions After Orthodontic Therapy: A Randomized Controlled Trial
Brief Title: White Spot Lesions Treatment in Orthodontic
Acronym: WSL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Riyadh Elm University (Other)
Responsible Party: Principal Investigator, Samira Fawaz M Algasn, Postgraduate Student, Riyadh Elm University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FPGRP/2023/780
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: White Spot Lesion
Keywords: Fixed orthodontic Appliances; White Spot Lesion; Fluoride Varnish; Casein Phosphopeptide-Amorphous Calcium Phosphate; Resin Infiltration; Laser Fluorescence
MeSH Terms: interventions — Sodium Fluoride; casein phosphopeptide-amorphous calcium phosphate nanocomplex

STUDY DESIGN:
Intervention Model Description: Once the FV has been applied, the examiners at Riyadh Elm University will do a visual inspection and take LF measurements (T2) on all the areas that were marked as WSL on the initial photos. The LF measurement will be carried out by the same inspectors who carried out the visual inspection.
  At the end of treatment for groups II, III, IV, a visual examination and LF measurements (T2) will be conducted by the same examiners. At the next inspection (after 3 months (T3)), LF measurements will be carried out on all areas that were marked as WSL on the original photos, whether they are still existing WSL areas or they will be changed to WSL free areas.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A web based research randomizer software will be used to generate a random sequence number to allocate the participants to different groups. The allocation will be kept concealed from patients and examiners using sequentially numbered identical containers containing experimental materials (remineralizing agents) to ensure the double blindness of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Fluoride Varnish (control) (Experimental): The study involves 22 patients with WSLs at Riyadh Elm University's dental clinics, who will undergo dental examinations and receive ICDAS codes. In group I, FV EnamelastTM will be applied to all teeth using compressed air and cotton rolls, leaving them to dry for one minute. Patients will be advised to avoid eating, drinking, or brushing for 3-4 hours after application.
  Interventions: Drug: 5% sodium fluoride
- Intensive Fluoride Varnish (Experimental): The study involves 22 patients with WSLs at Riyadh Elm University's dental clinics, who will undergo dental examinations and receive ICDAS codes. Patients in group II Intensive FV will be applied three times a week for a week (every two days).
  Interventions: Drug: Intensive 5% sodium fluoride
- Casein Phosphopeptide-Amorphous Calcium Phosphate (Experimental): The study involves 22 patients with WSLs at Riyadh Elm University's dental clinics, who will undergo dental examinations and receive ICDAS codes. Group III (CPP-ACP) uses Tooth Mousse® for 12 weeks, will be applied after daily brushing with traditional toothpaste, left intact for 180 seconds, and rinsed with distilled water.
  Interventions: Drug: Casein Phosphopeptide-Amorphous Calcium Phosphate
- Resin Infiltration (Experimental): The study involves 22 patients with WSLs at Riyadh Elm University's dental clinics, who will undergo dental examinations and receive ICDAS codes. Group IV uses ICON® resin infiltration, applying a 15% hydrochloric acid solution, rinsing with water, drying, and applying ICON-Dry. Excess resin is removed, and a light curing process is performed. The roughened enamel surface is polished using composite resin polish discs and cups.
  Interventions: Drug: Resin infiltration

INTERVENTIONS:
Drug: 5% sodium fluoride — a flavored xylitol-sweetened, 5% sodium fluoride in a resin carrier delivered in a 1.2 ml syringe or in a 0.4 ml unit, Ultradent, USA) will be applied on all teeth according to the manufacturer's instructions.
  Other Names: FV EnamelastTM
  Arms: Fluoride Varnish (control)
Drug: Intensive 5% sodium fluoride — Intensive FV will be applied three times a week for a week (every two days).
  Other Names: EnamelastTM
  Arms: Intensive Fluoride Varnish
Drug: Casein Phosphopeptide-Amorphous Calcium Phosphate — for 12 weeks. A thin layer from Tooth Mousse™ will be applied to the teeth after daily brushing with traditional toothpaste and left intact for 180 seconds before rinsing with distilled water
  Other Names: (CPP-ACP), Tooth Mousse® (MI Paste®) (GC Corporation, Tokyo, Japan)
  Arms: Casein Phosphopeptide-Amorphous Calcium Phosphate
Drug: Resin infiltration — resin infiltration will be applied as specified by the manufacturer.
  Other Names: ICON® (DMG, Hamburg, Germany)
  Arms: Resin Infiltration

SUMMARY:
The study aims to investigate the effectiveness of a new treatment for demineralized white spot lesions (WSLs) after fixed appliance therapy. The trial will consist of four parallel groups: control, Fluoride Varnish (FV), Casein Phosphopeptide-Amorphous Calcium Phosphate (CPP-ACP), and Resin Infiltration (RI) groups. Patients will be recruited from Riyadh Elm University's electronic record system and contacted by phone. They will be given an appointment to visit the dental clinic.

A total of 22 patients with WSLs will be selected for the study. Two examiners will perform dental examinations using a dental mirror and a ball-ended probe to code the WSL against the ICDAS system. The level of agreement between the two examiners will be assessed using reliability analysis, with an agreement level of above 80% considered.

Buccal WSLs will be defined as those that extend from the center of the buccal to either the mesial or distal surface. WSLs coded 3 or higher will be excluded from further examination and treated accordingly.

DETAILED DESCRIPTION:
Trial design The study will be conducted as a prospective clinical controlled trial with an experimental design, consisting of four parallel groups. Individuals who experienced the development of demineralized white spot lesions after undergoing fixed appliance therapy will be invited to participate in the study and will be assigned to one of the following groups: control group, Fluoride Varnish (FV) group, Casein Phosphopeptide-Amorphous Calcium Phosphate (CPP-ACP) group, or Resin Infiltration (RI) group.

Participants Patients will be recruited by navigating the electronic record system of Riyadh Elm University from 2023 files backward up to 2022, identifying patients who completed orthodontic treatment reaching up to the required sample size. Those patients will be contacted by phone call from the dental clinic of Riyadh Elm University official number, inviting them to participate in the current study. Patients will be given an appointment to visit the dental clinic at specific time. Before enrollment, every patient or parent/legal guardian of a patient younger than 18 years of age will receive an informational letter and verbal communication about the objectives and protocol of the study. All enrolled patients and/or their parents or legal guardians will be asked to provide a written informed consent following their initial approval. All patients who got treatment in Riyadh Elm University signed consents to share their information for research purposes will be enrolled in the study.

Calibration exercise A total of 22 patients with WSLs attending dental clinics of REU will be selected and two examiners will perform dental examinations using a dental mirror and a ball-ended probe on wet and dry debris-free teeth to code the WSL against the ICDAS system. Whenever in doubt regarding the coding of the WSLs, the third expert examiner decision will be considered final. The level of agreement with regard to the ICDAS codes between the two examiners will be assessed using reliability analysis and the agreement level of above 80% will be considered.

Two examiners will perform dental examinations using a dental mirror and a ball-ended probe on wet and dry debris-free teeth. Each WSL will be identified by visual inspection of mesiobuccal, buccal, or distobuccal tooth surfaces and recorded. An ICDAS code will be assigned to each WSL. A digital photograph will be taken by keeping 45 cm distance between subject and camera. The digital image of WS can be captured with a digital camera (Canon EOS 2000D (NIS) DSLR Camera 18 - 55 mm NIS Lens) held almost perpendicular to the buccal surface. Light is supplied by a flash mounted around lens. The camera system setup was adjusted as follows; the quality of image is Fine, ISO is 200, and white balance is speed light mode. Moreover, dental status of the participants also recorded.

Buccal WSLs will be defined as those that extend from the center of the buccal to either the mesial surface or the distal surface. WSLs that will be coded 3 (denoted by localized enamel breakdown caused by caries without the presence of dentin and underlying shadow), or higher (denoted by the presence of underlying dark shadow caused by dentin, whether enamel-depleting or not, to a large distinct cavity containing visible dentin), in accordance with ICDAS reference, are excluded from further examination and will be appropriately treated.

Following the determination of the 0 LF value for each tooth on a healthy surface, the maximum LF value for each WSL coded tooth (either 1 or 2) will be determined using a DIAGNODent flat tip (KaVo dental, GmbH, Biberach, Germany). Measurements will be done according to the manufacturer's instructions. Each tooth will be dried for 5 seconds, and the tip will be pointed in the opposite direction from the examination area. The measurement will be done using the DIAGNOdent Scale; values 0±13: no caries, values 14±20: enamel caries and values >20: dentinal caries. (Lussi et al., 2001).

Eligibility criteria for participants Inclusion criteria

1. Post orthodontic patients with one WSLs on buccal surface of tooth with ICDAS Code 1 or 2.
2. Agreeing to participate in the study by singing the study informed consent.
3. For younger patients parents agree to provide consent for child participation in the study.

Exclusion criteria

1. Developmental defects of dental hard tissue
2. Patients who have systemic disease or under medications that usually cause an increased risk of oral caries.
3. Patients who are allergic to Fluoride varnish, CPP-ACP and resin infiltration. Study settings Data will be collected from orthodontic clinics of Namouthajya and Muneseya hospitals at Riyadh Elm University, Riyadh, Saudi Arabia.

Intervention In group I (Control group): FV EnamelastTM (a flavored xylitol-sweetened, 5% sodium fluoride in a resin carrier delivered in a 1.2 ml syringe or in a 0.4 ml unit, Ultradent, USA) will be applied on all teeth according to the manufacturer's instructions: compressed air and cotton rolls will be used to dry the teeth. A mini brush will be used to apply varnish to all teeth surfaces. The varnish will be left to dry for one minute. Patients should avoid eating, drinking, or brushing for a period of 3-4 hours following the application of varnish. In the test groups (group II): Intensive FV will be applied three times a week for a week (every two days). For group III: (CPP-ACP), Tooth Mousse® (MI Paste®) (GC Corporation, Tokyo, Japan) for 12 weeks. A thin layer from Tooth Mousse™ will be applied to the teeth after daily brushing with traditional toothpaste and left intact for 180 seconds before rinsing with distilled water (Thierens et al., 2019). For group IV: ICON® (DMG, Hamburg, Germany) resin infiltration will be applied as specified by the manufacturer: the 15% hydrochloric acid (HCL) solution will be sprayed for 2 minutes, followed by rinsing with water for 30 seconds and drying. Application of ICON-Dry (Ethanol) for 30 seconds, followed by air drying. Subsequently, ICON-Infiltration will be applied to the tooth surface and left for 3 minutes. The excess resin will be removed using a cotton roll, followed by a light curing process lasting for 40 seconds. Finally, the enamel surface that has been roughened will be polished with composite resin polish discs and polish cups.

ELIGIBILITY:
Inclusion Criteria:

1. Post orthodontic patients with one WSLs on buccal surface of tooth with ICDAS Code 1 or 2.
2. Agreeing to participate in the study by singing the study informed consent.
3. For younger patients parents agree to provide consent for child participation in the study.

Exclusion Criteria:

1. Developmental defects of dental hard tissue
2. Patients who have systemic disease or under medications that usually cause an increased risk of oral caries.
3. Patients who are allergic to Fluoride varnish, CPP-ACP and resin infiltration.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Change in mineral contents of enamel | Baseline pre-treatment (T1), immediately post-treatment (T2), and three months post-treatment (T3)
  The maximum light fluorescence value for each tooth with a white spot lesion will be determined using a DIAGNODent flat tip, following manufacturer's instructions. The DIAGNOdent scale will be used to measure the mineral content of enamel, with values ranging from 0 to 20.

CONTACTS AND LOCATIONS:
Overall Officials: Samira Algasn, BDS, Principal Investigator — Riyadh Elm University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boersma JG, van der Veen MH, Lagerweij MD, Bokhout B, Prahl-Andersen B. Caries prevalence measured with QLF after treatment with fixed orthodontic appliances: influencing factors. Caries Res. 2005 Jan-Feb;39(1):41-7. doi: 10.1159/000081655. PMID 15591733
- [Background] Ferreira JM, Silva MF, Oliveira AF, Sampaio FC. Evaluation of different methods for monitoring incipient carious lesions in smooth surfaces under fluoride varnish therapy. Int J Paediatr Dent. 2008 Jul;18(4):300-5. doi: 10.1111/j.1365-263X.2007.00879.x. PMID 18554336
- [Background] Lussi A, Megert B, Longbottom C, Reich E, Francescut P. Clinical performance of a laser fluorescence device for detection of occlusal caries lesions. Eur J Oral Sci. 2001 Feb;109(1):14-9. doi: 10.1034/j.1600-0722.2001.109001014.x. PMID 11330928
- [Background] Makhija SK, Bader JD, Shugars DA, Litaker MS, Nagarkar S, Gordan VV, Rindal DB, Pihlstrom DJ, Mungia R, Meyerowitz C, Gilbert GH; National Dental Practice-Based Research Network (PBRN) Collaborative Group. Influence of 2 caries-detecting devices on clinical decision making and lesion depth for suspicious occlusal lesions: A randomized trial from The National Dental Practice-Based Research Network. J Am Dent Assoc. 2018 Apr;149(4):299-307.e1. doi: 10.1016/j.adaj.2017.11.001. Epub 2018 Feb 21. PMID 29475554
- [Background] Melrose CA, Appleton J, Lovius BB. A scanning electron microscopic study of early enamel caries formed in vivo beneath orthodontic bands. Br J Orthod. 1996 Feb;23(1):43-7. doi: 10.1179/bjo.23.1.43. PMID 8652497
- [Background] Migliorati M, Isaia L, Cassaro A, Rivetti A, Silvestrini-Biavati F, Gastaldo L, Piccardo I, Dalessandri D, Silvestrini-Biavati A. Efficacy of professional hygiene and prophylaxis on preventing plaque increase in orthodontic patients with multibracket appliances: a systematic review. Eur J Orthod. 2015 Jun;37(3):297-307. doi: 10.1093/ejo/cju044. Epub 2014 Sep 22. PMID 25246605
- [Result] Aljehani A, Yousif MA, Angmar-Mansson B, Shi XQ. Longitudinal quantification of incipient carious lesions in postorthodontic patients using a fluorescence method. Eur J Oral Sci. 2006 Oct;114(5):430-4. doi: 10.1111/j.1600-0722.2006.00395.x. PMID 17026510
- [Result] Eckstein A, Helms HJ, Knosel M. Camouflage effects following resin infiltration of postorthodontic white-spot lesions in vivo: One-year follow-up. Angle Orthod. 2015 May;85(3):374-80. doi: 10.2319/050914-334.1. Epub 2014 Aug 15. PMID 25126675
- [Result] Kau CH, Wang J, Palombini A, Abou-Kheir N, Christou T. Effect of fluoride dentifrices on white spot lesions during orthodontic treatment: A randomized trial. Angle Orthod. 2019 May;89(3):365-371. doi: 10.2319/051818-371.1. Epub 2019 Feb 5. PMID 30719933
- [Result] Llena C, Leyda AM, Forner L. CPP-ACP and CPP-ACFP versus fluoride varnish in remineralisation of early caries lesions. A prospective study. Eur J Paediatr Dent. 2015 Sep;16(3):181-6. PMID 26418918
- [Result] Meyer-Lueckel H, Paris S. Progression of artificial enamel caries lesions after infiltration with experimental light curing resins. Caries Res. 2008;42(2):117-24. doi: 10.1159/000118631. Epub 2008 Feb 28. PMID 18305389
- [Result] Nascimento PL, Fernandes MT, Figueiredo FE, Faria-E-Silva AL. Fluoride-Releasing Materials to Prevent White Spot Lesions around Orthodontic Brackets: A Systematic Review. Braz Dent J. 2016 Jan-Feb;27(1):101-7. doi: 10.1590/0103-6440201600482. PMID 27007355
- [Result] Sonesson M, Brechter A, Lindman R, Abdulraheem S, Twetman S. Fluoride varnish for white spot lesion prevention during orthodontic treatment: results of a randomized controlled trial 1 year after debonding. Eur J Orthod. 2021 Aug 3;43(4):473-477. doi: 10.1093/ejo/cjaa055. PMID 33009565
- See also: CPP-ACP and CPP-ACFP versus fluoride varnish in remineralisation of early caries lesions. A prospective study — https://pubmed.ncbi.nlm.nih.gov/26418918/